CLINICAL TRIAL: NCT01514240
Title: A Multicentre, Double-blind, Randomised, Parallel-group, Phase III Study to Assess Efficacy and Safety of D9421-C 9 mg Versus Mesalazine 3 g in Patients With Active Crohn's Disease (CD) in Japan
Brief Title: Phase III Study of D9421-C 9 mg in Patients With Active Crohn's Disease in Japan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D9423C00001
Record Dates: First submitted 2012-01-10; First posted 2012-01-23 (Estimated); Results first posted 2016-10-31 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-09

CONDITIONS: Crohn's Disease
Keywords: mild to moderate active Crohn's disease; affecting ileum; ileocecal region; ascending colon; score of 180-400 on the CDAI
MeSH Terms: conditions — Crohn Disease | interventions — Mesalamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- D9421-C (Experimental): D9421-C 9 mg once daily
  Interventions: Drug: D9421-C capsule 3 mg
- Mesalazine (Active Comparator): Mesalazine 1 g three times a day
  Interventions: Drug: Mesalazine tablets

INTERVENTIONS:
Drug: D9421-C capsule 3 mg — Patients randomised to D9421-C 9 mg will take 3 capsules of D9421-C capsule 3 mg once daily before breakfast and 4 tablets of Mesalazine tablets placebo three times a day after each meal for 8 weeks.
  Arms: D9421-C
Drug: Mesalazine tablets — Patients randomised to Mesalazine 3 g will take 3 capsules of D9421-C capsule placebo once daily before breakfast and 4 tablets of Mesalazine tablets 250 mg three times a day after each meal for 8 weeks.
  Arms: Mesalazine

SUMMARY:
The purpose of this study is to evaluate the clinical efficacy of D9421-C 9 mg once daily compared to Mesalazine 1 g three times a day to patients with mild to moderate active Crohn's disease affecting ileum, ileocecal region and/or ascending colon as defined by a score of 180-400 on the Crohn's Disease Activity Index (CDAI) by assessment of the remission after 8-week treatment defined by a CDAI score of ≤ 150.

DETAILED DESCRIPTION:
A multicentre, double-blind, randomised, parallel-group, Phase III study to assess efficacy and safety of D9421-C 9 mg versus Mesalazine 3 g in patients with active Crohn's Disease (CD) in Japan

ELIGIBILITY:
Inclusion Criteria:

* 15 years of age or older
* Main active disease of the ileal, ileocecal region, and/or ascending colon - - If treated with partial nutrition treatment (≤1200 kcal/day) or if treated with azathioprine (≤2.0 mg/kg/day) or 6-mercaptopurine (≤1.2 mg/kg/day), prior to randomisation until the study completion or discontinuation
* Ability to read, write and to fill a diary card and HRQL questionnaire Having mild to moderate active Crohn's disease, defined as CDAI score of 180-400 at baseline

Exclusion Criteria:

* Patient with CD lesion or status which may affect the evaluation of the efficacy (e.g. lesion only in the upper G-I, active anorectal lesion, abscess formation, stenosis, fistulae, ostomy, short bowel or other uncontrolled concomitant disease)
* Patient who need any concomitant treatment for CD that may affect the assessment for efficacy of the study drug
* Patient who need any medication which is prohibited due to suspected influence to metabolism of the study drug
* Patient who is judged to be inadequate to participate in this study from the safety point of view Patient with well-founded doubt about protocol violation

Ages: 15 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2012-02; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Toshifumi Hibi, Professor, Chairman, Principal Investigator — Department of Internal Medicine, Keio University School of Medicine
Locations (25):
- Japan (25):
  - Research Site, Chikushino-shi
  - Research Site, Fukuoka
  - Research Site, Fukuyama-shi
  - Research Site, Hirosaki-shi
  - Research Site, Hiroshima
  - Research Site, Kagoshima
  - Research Site, Kitakyushu-shi
  - Research Site, Koshigaya-shi
  - Research Site, Kurume-shi
  - Research Site, Kyoto
  - Research Site, Nagakute-shi
  - Research Site, Nagoya
  - Research Site, Nishinomiya-shi
  - Research Site, Okayama
  - Research Site, Omura-shi
  - Research Site, Osaka
  - Research Site, Ōita
  - Research Site, Sakura
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Shinjyuku-ku
  - Research Site, Suginami-ku
  - Research Site, Suita-shi
  - Research Site, Toyoake-shi
  - Research Site, Toyota-shi

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled on 08 February 2012. Last subject last visit on 08 September 2014.
Pre-assignment Details: Out of 123 enrolled subjects, 112 subjects were randomised and 11 subjects were not randomised. The reasons of no randomisation were 'Eligibility criteria not met' (9 subjects) and 'Adverse event' (2 subjects).
Groups:
- D9421-C 9mg + Mesalazine Placebo: Patients randomised to D9421-C 9 mg took 3 capsules of D9421-C capsule 3 mg once daily before breakfast and 4 tablets of Mesalazine tablets placebo three times a day after each meal for 8 weeks.
- Mesalazine 3g + D9421-C Placebo: Patients randomised to Mesalazine 3 g took 3 capsules of D9421-C capsule placebo once daily before breakfast and 4 tablets of Mesalazine tablets 250 mg three times a day after each meal for 8 weeks.
Period: Overall Study
Arm/Group | D9421-C 9mg + Mesalazine Placebo | Mesalazine 3g + D9421-C Placebo
Started | 56 | 56
Completed | 50 | 45
Not Completed | 6 | 11
Not completed — Adverse Event | 4 | 4
Not completed — Subject Decision | 2 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | D9421-C 9mg + Mesalazine Placebo | Mesalazine 3g + D9421-C Placebo | Total
Number analyzed (Participants) | 56 | 56 | 112
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.1 (13.43) [16 to 77] | 35.8 (10.71) [19 to 64] | 36.9 (12.15) [16 to 77]
Age, Customized [Number; unit: Participants]
  <30 Years | 19 | 20 | 39
  >=30 Years | 37 | 36 | 73
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 13 | 32
  Male | 37 | 43 | 80
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 56 | 55 | 111
  Black/African American | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Remission After 8-week of Treatment
Description: For the primary efficacy variable "Remission after 8 weeks of treatment", Crohn's Disease Activity Index CDAI scores was used to determine the patient's response. Remission for this study is defined as a CDAI score of ≤150. A patient who drops out without any remission before week 8 was considered as a nonresponder (no remission) for this analysis. A patient who drops out before Week 8, but was in remission at the time of dropout, was considered in remission after dropout in this analysis.
Time Frame: 8 Week
Population: All randomised patients who take the investigational products at least once and have data in the treatment period
Measure: Number; unit: Participants
Arm/Group | D9421-C 9mg + Mesalazine Placebo | Mesalazine 3g + D9421-C Placebo
Number analyzed (Participants) | 56 | 56
Participants | 17 | 14
Statistical Analysis 1: Comparison: D9421-C 9mg + Mesalazine Placebo vs Mesalazine 3g + D9421-C Placebo; The primary objective of this study was to determine non-inferiority in the differences in remission rates at Week 8 for D9421-C 9 mg as compared to Mesalazine 3 g; Test type: Non-Inferiority or Equivalence — A 2-sided 90% CI for the observed difference in the primary outcome measure (remission rate) between the D9421-C 9mg group and the Mesalazine 3 g group was calculated at week 8 using the Newcombe-Wilson score method without continuity correction. Noninferiority was concluded if the lower limit of the 90% CI was higher than -10% in FAS Population; p = 0.526, Chi-squared; Difference of proportion = 5.4, 90% CI 2-sided [-8.49 to 18.94]

2. Secondary Outcome: Remission After 2-week of Treatment
Description: For the secondary efficacy variable "Remission after 2 weeks of treatment", Crohn's Disease Activity Index CDAI scores was used to determine the patient's response. Remission for this study is defined as a CDAI score of ≤150.
Time Frame: 2 Week
Population: All randomised patients who take the investigational products at least once and have data in the treatment period
Measure: Number; unit: Participants
Arm/Group | D9421-C 9mg + Mesalazine Placebo | Mesalazine 3g + D9421-C Placebo
Number analyzed (Participants) | 56 | 56
Participants | 7 | 6
Statistical Analysis 1: Comparison: D9421-C 9mg + Mesalazine Placebo vs Mesalazine 3g + D9421-C Placebo; Test type: Superiority or Other; p = 0.768, Chi-squared; Difference of proportion = 1.8, 90% CI 2-sided [-8.54 to 12.15] — Differences in remission rate at Week 2 between D9421-C 9 mg and Mesalazine 3 g along with their 2-sided 90% CIs calculated by the Newcombe-Wilson score method without continuity correction

3. Secondary Outcome: Remission After 4-week of Treatment
Description: For the secondary efficacy variable "Remission after 4 weeks of treatment", Crohn's Disease Activity Index CDAI scores was used to determine the patient's response. Remission for this study is defined as a CDAI score of ≤150.
Time Frame: 4 Week
Population: All randomised patients who take the investigational products at least once and have data in the treatment period
Measure: Number; unit: Participants
Arm/Group | D9421-C 9mg + Mesalazine Placebo | Mesalazine 3g + D9421-C Placebo
Number analyzed (Participants) | 56 | 56
Participants | 12 | 7
Statistical Analysis 1: Comparison: D9421-C 9mg + Mesalazine Placebo vs Mesalazine 3g + D9421-C Placebo; Test type: Superiority or Other; p = 0.208, Chi-squared; Difference of proportion = 8.9, 90% CI 2-sided [-2.87 to 20.58] — Differences in remission rate at Week 4 between D9421-C 9 mg and Mesalazine 3 g along with their 2-sided 90% CIs calculated by the Newcombe-Wilson score method without continuity correction

4. Secondary Outcome: Change in Observed CDAI Scores From Baseline to Weeks 2
Description: Crohn's Disease Activity Index (CDAI) score is calculated based on the data collected in the diary card. The total CDAI score ranges from 0 to approximately 600, a higher scores indicating more severe disease. The target population of total CDAI score 180 to 400 is defined mild to modarate active Crohn's disease. Total CDAI score 150 less or equal is evaluated as a remission.
  Patients are asked to fill the following items in the diary card (from the morning in preceding day to the morning in current day). (1) Number of liquid or very soft stools (2) Abdominal pain rating (none, mild, moderate, severe) (3) General well-being (generally well, slightly under par, poor, very poor, terrible) (4) Body temperature (if a patient feels fever) (5) Intake of loperamide or other opiates for diarrhoea. The data for the calculation of CDAI score in diary card is then transcribed by the investigator(s) into the eCRFs at each clinical visit.
Time Frame: 2 Week
Population: All randomised patients who take the investigational products at least once and have data in the treatment period. However, the patients with both baseline and week 2 data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | D9421-C 9mg + Mesalazine Placebo | Mesalazine 3g + D9421-C Placebo
Number analyzed (Participants) | 53 | 53
Scores on a scale | -38.5 (8.91) | -15.7 (7.66)
Statistical Analysis 1: Comparison: D9421-C 9mg + Mesalazine Placebo vs Mesalazine 3g + D9421-C Placebo; Test type: Superiority or Other; p = 0.058, Mixed Models Analysis; LS mean difference between group = -22.8, 90% CI 2-sided [-42.55 to -3.09], Standard Error of Mean 11.89 — The analysis using a MMRM analysis including a covariate of the corresponding score at baseline,fixed effects of time (as a categorical factor) and treatment and interaction between time and treatment group

5. Secondary Outcome: Change in Observed CDAI Scores From Baseline to Weeks 4
Description: as for outcome 4
Time Frame: 4 Week
Population: All randomised patients who take the investigational products at least once and have data in the treatment period. However, the patients with both baseline and week 4 data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | D9421-C 9mg + Mesalazine Placebo | Mesalazine 3g + D9421-C Placebo
Number analyzed (Participants) | 55 | 50
Scores on a scale | -58.7 (9.44) | -28.7 (7.29)
Statistical Analysis 1: Comparison: D9421-C 9mg + Mesalazine Placebo vs Mesalazine 3g + D9421-C Placebo; Test type: Superiority or Other; p = 0.014, Mixed Models Analysis; LS mean difference between group = -30.0, 90% CI 2-sided [-49.95 to -9.96], Standard Error of Mean 12.05 — [estimate comment as in outcome 4, analysis 1]

6. Secondary Outcome: Change in Observed CDAI Scores From Baseline to Weeks 8
Description: as for outcome 4
Time Frame: 8 Week
Population: All randomised patients who take the investigational products at least once and have data in the treatment period. However, the patients with both baseline and week 8 data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | D9421-C 9mg + Mesalazine Placebo | Mesalazine 3g + D9421-C Placebo
Number analyzed (Participants) | 51 | 45
Scores on a scale | -67.0 (11.17) | -45.7 (9.11)
Statistical Analysis 1: Comparison: D9421-C 9mg + Mesalazine Placebo vs Mesalazine 3g + D9421-C Placebo; Test type: Superiority or Other; p = 0.144, Mixed Models Analysis; LS mean difference between group = -21.4, 90% CI 2-sided [-45.47 to 2.74], Standard Error of Mean 14.53 — [estimate comment as in outcome 4, analysis 1]

7. Secondary Outcome: Cumulative Remission Rate at Week 2
Description: Remission rate is defined as CDAI score of less than or equal to 150. Cumulative remission rate at Week 2 is obtained by Kaplan-Meier (KM) estimates.
Time Frame: 2 Week
Population: All randomised patients who take the investigational products at least once and have data in the treatment period
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | D9421-C 9mg + Mesalazine Placebo | Mesalazine 3g + D9421-C Placebo
Number analyzed (Participants) | 56 | 56
Percentage of participants | 12.5 [5.23 to 19.77] | 10.7 [3.92 to 17.51]

8. Secondary Outcome: Cumulative Remission Rate at Week 4
Description: Remission rate is defined as CDAI score of less than or equal to 150. Cumulative remission rate at Week 4 is obtained by Kaplan-Meier (KM) estimates.
Time Frame: 4 Week
Population: All randomised patients who take the investigational products at least once and have data in the treatment period
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | D9421-C 9mg + Mesalazine Placebo | Mesalazine 3g + D9421-C Placebo
Number analyzed (Participants) | 56 | 56
Percentage of participants | 25.0 [15.48 to 34.52] | 17.9 [9.44 to 26.28]

9. Secondary Outcome: Cumulative Remission Rate at Week 8
Description: Remission rate is defined as CDAI score of less than or equal to 150. Cumulative remission rate at Week 8 is obtained by Kaplan-Meier (KM) estimates.
Time Frame: 8 Week
Population: All randomised patients who take the investigational products at least once and have data in the treatment period
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | D9421-C 9mg + Mesalazine Placebo | Mesalazine 3g + D9421-C Placebo
Number analyzed (Participants) | 56 | 56
Percentage of participants | 37.5 [26.86 to 48.14] | 30.4 [20.25 to 40.46]

10. Secondary Outcome: Clinical Improvement Rates (Decrease in CDAI Score From Baseline of at Least 70 Points) at Weeks 2
Description: Clinical improvement is defined as CDAI score of <=150 or a decrease in CDAI score from baseline of at least 70 points.
Time Frame: 2 Week
Population: All randomised patients who take the investigational products at least once and have data in the treatment period.
Measure: Number; unit: Participants
Arm/Group | D9421-C 9mg + Mesalazine Placebo | Mesalazine 3g + D9421-C Placebo
Number analyzed (Participants) | 56 | 56
Participants | 19 (9.07) | 11 (7.46)
Statistical Analysis 1: Comparison: D9421-C 9mg + Mesalazine Placebo vs Mesalazine 3g + D9421-C Placebo; Test type: Superiority or Other; Difference of proportions = 14.3, 90% CI 2-sided [0.50 to 27.40] — 90% CI calculated using the Newcombe-Wilson score method without continuity corrections

11. Secondary Outcome: Clinical Improvement Rates (Decrease in CDAI Score From Baseline of at Least 70 Points) at Weeks 4
Description: Clinical improvement is defined as CDAI score of <=150 or a decrease in CDAI score from baseline of at least 70 points.
Time Frame: 4 Week
Population: All randomised patients who take the investigational products at least once and have data in the treatment period.
Measure: Number; unit: Participants
Arm/Group | D9421-C 9mg + Mesalazine Placebo | Mesalazine 3g + D9421-C Placebo
Number analyzed (Participants) | 56 | 56
Participants | 22 (9.07) | 13 (7.46)
Statistical Analysis 1: Comparison: D9421-C 9mg + Mesalazine Placebo vs Mesalazine 3g + D9421-C Placebo; Test type: Superiority or Other; Difference of proportions = 16.1, 90% CI 2-sided [1.66 to 29.61] — 90% CI calculated using the Newcombe-Wilson score method without continuity corrections

12. Secondary Outcome: Clinical Improvement Rates (Decrease in CDAI Score From Baseline of at Least 70 Points) at Weeks 8
Description: Clinical improvement is defined as CDAI score of <=150 or a decrease in CDAI score from baseline of at least 70 points.
Time Frame: 8 Week
Population: All randomised patients who take the investigational products at least once and have data in the treatment period.
Measure: Number; unit: Participants
Arm/Group | D9421-C 9mg + Mesalazine Placebo | Mesalazine 3g + D9421-C Placebo
Number analyzed (Participants) | 56 | 56
Participants | 27 (9.07) | 18 (7.46)
Statistical Analysis 1: Comparison: D9421-C 9mg + Mesalazine Placebo vs Mesalazine 3g + D9421-C Placebo; Test type: Superiority or Other; Difference of proportions = 16.1, 90% CI 2-sided [0.85 to 30.29] — 90% CI calculated using the Newcombe-Wilson score method without continuity corrections

13. Secondary Outcome: Clinical Improvement Rates (Decrease in CDAI Score From Baseline of at Least 100 Points) at Weeks 2
Description: Clinical improvement is defined as CDAI score of <=150 or a decrease in CDAI score from baseline of at least 100 points.
Time Frame: 2 Week
Population: All randomised patients who take the investigational products at least once and have data in the treatment period.
Measure: Number; unit: Participants
Arm/Group | D9421-C 9mg + Mesalazine Placebo | Mesalazine 3g + D9421-C Placebo
Number analyzed (Participants) | 56 | 56
Participants | 14 (9.07) | 10 (7.46)
Statistical Analysis 1: Comparison: D9421-C 9mg + Mesalazine Placebo vs Mesalazine 3g + D9421-C Placebo; Test type: Superiority or Other; Difference of proportions = 7.1, 90% CI 2-sided [-5.67 to 19.71] — 90% CI calculated using the Newcombe-Wilson score method without continuity corrections

14. Secondary Outcome: Clinical Improvement Rates (Decrease in CDAI Score From Baseline of at Least 100 Points) at Weeks 4
Description: Clinical improvement is defined as CDAI score of <=150 or a decrease in CDAI score from baseline of at least 100 points.
Time Frame: 4 Week
Population: All randomised patients who take the investigational products at least once and have data in the treatment period.
Measure: Number; unit: Participants
Arm/Group | D9421-C 9mg + Mesalazine Placebo | Mesalazine 3g + D9421-C Placebo
Number analyzed (Participants) | 56 | 56
Participants | 19 (9.07) | 11 (7.46)
Statistical Analysis 1: Comparison: D9421-C 9mg + Mesalazine Placebo vs Mesalazine 3g + D9421-C Placebo; Test type: Superiority or Other; Difference of proportions = 14.3, 90% CI 2-sided [0.50 to 27.40] — 90% CI calculated using the Newcombe-Wilson score method without continuity corrections

15. Secondary Outcome: Clinical Improvement Rates (Decrease in CDAI Score From Baseline of at Least 100 Points) at Weeks 8
Description: Clinical improvement is defined as CDAI score of <=150 or a decrease in CDAI score from baseline of at least 100 points.
Time Frame: 8 Week
Population: All randomised patients who take the investigational products at least once and have data in the treatment period.
Measure: Number; unit: Participants
Arm/Group | D9421-C 9mg + Mesalazine Placebo | Mesalazine 3g + D9421-C Placebo
Number analyzed (Participants) | 56 | 56
Participants | 24 (9.07) | 17 (7.46)
Statistical Analysis 1: Comparison: D9421-C 9mg + Mesalazine Placebo vs Mesalazine 3g + D9421-C Placebo; Test type: Superiority or Other; Difference of proportions = 12.5, 90% CI 2-sided [-2.44 to 26.68] — 90% CI calculated using the Newcombe-Wilson score method without continuity corrections

16. Secondary Outcome: Change in Total IBDQ Scores From Baseline to Weeks 2
Description: The Inflammatory Bowel Disease Questionnaire (IBDQ) is a standard measure of HRQL in Crohn's disease patients (Guyatt G et al 1989). The validated Japanese version of the IBDQ was used in this study (Hashimoto H et al 2003). The IBDQ contains 32 questions; each with seven possible answers ranging from 1 to 7, where 7 is the most favourable. Ten questions are related to bowel symptoms, five to systemic symptoms, twelve to emotional function, and five to social function. The corresponding answers will be added to form four subscores and a total score: bowel function score (10 - 70), systemic symptom score (5 - 35), emotional function score (12 - 84), social function score (5 - 35) and the total score (32 - 224), with higher scores indicating more favorable outcome.
Time Frame: 2 Week
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | D9421-C 9mg + Mesalazine Placebo | Mesalazine 3g + D9421-C Placebo
Number analyzed (Participants) | 56 | 54
Scores on a scale | 16.2 (2.30) | 5.7 (2.41)
Statistical Analysis 1: Comparison: D9421-C 9mg + Mesalazine Placebo vs Mesalazine 3g + D9421-C Placebo; Test type: Superiority or Other; LS mean difference between group = 10.5, 90% CI 2-sided [4.86 to 16.14], Standard Error of Mean 3.40 — [estimate comment as in outcome 4, analysis 1]

17. Secondary Outcome: Change in Total IBDQ Scores From Baseline to Weeks 4
Description: as for outcome 16
Time Frame: 4 Week
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | D9421-C 9mg + Mesalazine Placebo | Mesalazine 3g + D9421-C Placebo
Number analyzed (Participants) | 55 | 50
Scores on a scale | 19.4 (3.03) | 6.8 (2.44)
Statistical Analysis 1: Comparison: D9421-C 9mg + Mesalazine Placebo vs Mesalazine 3g + D9421-C Placebo; Test type: Superiority or Other; LS mean difference between group = 12.6, 90% CI 2-sided [6.07 to 19.11], Standard Error of Mean 3.93 — [estimate comment as in outcome 4, analysis 1]

18. Secondary Outcome: Change in Total IBDQ Scores From Baseline to Weeks 8
Description: as for outcome 16
Time Frame: 8 Week
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | D9421-C 9mg + Mesalazine Placebo | Mesalazine 3g + D9421-C Placebo
Number analyzed (Participants) | 51 | 45
Scores on a scale | 18.3 (2.93) | 5.8 (3.16)
Statistical Analysis 1: Comparison: D9421-C 9mg + Mesalazine Placebo vs Mesalazine 3g + D9421-C Placebo; Test type: Superiority or Other; LS mean difference between group = 12.6, 90% CI 2-sided [5.40 to 19.72], Standard Error of Mean 4.31 — [estimate comment as in outcome 4, analysis 1]

19. Secondary Outcome: Change in Total IBDQ Scores From Baseline to Weeks 10
Description: as for outcome 16
Time Frame: 10 Week
Population: All randomised patients who take the investigational products at least once and have data in the treatment period. However, the patients with both baseline and week 10 data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | D9421-C 9mg + Mesalazine Placebo | Mesalazine 3g + D9421-C Placebo
Number analyzed (Participants) | 50 | 45
Scores on a scale | 21.1 (3.11) | 7.1 (2.96)
Statistical Analysis 1: Comparison: D9421-C 9mg + Mesalazine Placebo vs Mesalazine 3g + D9421-C Placebo; Test type: Superiority or Other; LS mean difference between group = 14.1, 90% CI 2-sided [6.90 to 21.23], Standard Error of Mean 4.32 — [estimate comment as in outcome 4, analysis 1]

20. Secondary Outcome: Change in IBDQ Scores From Baseline to Weeks 2 - Bowel Function
Description: as for outcome 16
Time Frame: 2 Week
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | D9421-C 9mg + Mesalazine Placebo | Mesalazine 3g + D9421-C Placebo
Number analyzed (Participants) | 56 | 54
Scores on a scale | 6.1 (0.77) | 2.7 (0.82)
Statistical Analysis 1: Comparison: D9421-C 9mg + Mesalazine Placebo vs Mesalazine 3g + D9421-C Placebo; Test type: Superiority or Other; LS mean difference between group = 3.4, 90% CI 2-sided [1.49 to 5.29], Standard Error of Mean 1.14 — [estimate comment as in outcome 4, analysis 1]

21. Secondary Outcome: Change in IBDQ Scores From Baseline to Weeks 4 - Bowel Function
Description: as for outcome 16
Time Frame: 4 Week
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | D9421-C 9mg + Mesalazine Placebo | Mesalazine 3g + D9421-C Placebo
Number analyzed (Participants) | 55 | 50
Scores on a scale | 6.6 (0.99) | 2.8 (0.84)
Statistical Analysis 1: Comparison: D9421-C 9mg + Mesalazine Placebo vs Mesalazine 3g + D9421-C Placebo; Test type: Superiority or Other; LS mean difference between group = 3.8, 90% CI 2-sided [1.64 to 5.97], Standard Error of Mean 1.31 — [estimate comment as in outcome 4, analysis 1]

22. Secondary Outcome: Change in IBDQ Scores From Baseline to Weeks 8 - Bowel Function
Description: as for outcome 16
Time Frame: 8 Week
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | D9421-C 9mg + Mesalazine Placebo | Mesalazine 3g + D9421-C Placebo
Number analyzed (Participants) | 51 | 45
Scores on a scale | 6.5 (1.04) | 2.4 (1.11)
Statistical Analysis 1: Comparison: D9421-C 9mg + Mesalazine Placebo vs Mesalazine 3g + D9421-C Placebo; Test type: Superiority or Other; LS mean difference between group = 4.1, 90% CI 2-sided [1.58 to 6.64], Standard Error of Mean 1.53 — [estimate comment as in outcome 4, analysis 1]

23. Secondary Outcome: Change in IBDQ Scores From Baseline to Weeks 10 - Bowel Function
Description: as for outcome 16
Time Frame: 10 Week
Population: as for outcome 19
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | D9421-C 9mg + Mesalazine Placebo | Mesalazine 3g + D9421-C Placebo
Number analyzed (Participants) | 50 | 45
Scores on a scale | 6.9 (1.08) | 3.6 (0.98)
Statistical Analysis 1: Comparison: D9421-C 9mg + Mesalazine Placebo vs Mesalazine 3g + D9421-C Placebo; Test type: Superiority or Other; LS mean difference between group = 3.3, 90% CI 2-sided [0.90 to 5.76], Standard Error of Mean 1.47 — [estimate comment as in outcome 4, analysis 1]

24. Secondary Outcome: Change in IBDQ Scores From Baseline to Weeks 2 - Systemic Symptom
Description: as for outcome 16
Time Frame: 2 Week
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | D9421-C 9mg + Mesalazine Placebo | Mesalazine 3g + D9421-C Placebo
Number analyzed (Participants) | 56 | 54
Scores on a scale | 3.0 (0.49) | 1.0 (0.48)
Statistical Analysis 1: Comparison: D9421-C 9mg + Mesalazine Placebo vs Mesalazine 3g + D9421-C Placebo; Test type: Superiority or Other; LS mean difference between group = 2.0, 90% CI 2-sided [0.89 to 3.17], Standard Error of Mean 0.69 — [estimate comment as in outcome 4, analysis 1]

25. Secondary Outcome: Change in IBDQ Scores From Baseline to Weeks 4 - Systemic Symptom
Description: as for outcome 16
Time Frame: 4 Week
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | D9421-C 9mg + Mesalazine Placebo | Mesalazine 3g + D9421-C Placebo
Number analyzed (Participants) | 55 | 50
Scores on a scale | 3.3 (0.57) | 1.3 (0.47)
Statistical Analysis 1: Comparison: D9421-C 9mg + Mesalazine Placebo vs Mesalazine 3g + D9421-C Placebo; Test type: Superiority or Other; LS mean difference between group = 2.0, 90% CI 2-sided [0.73 to 3.19], Standard Error of Mean 0.74 — [estimate comment as in outcome 4, analysis 1]

26. Secondary Outcome: Change in IBDQ Scores From Baseline to Weeks 8 - Systemic Symptom
Description: as for outcome 16
Time Frame: 8 Week
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | D9421-C 9mg + Mesalazine Placebo | Mesalazine 3g + D9421-C Placebo
Number analyzed (Participants) | 51 | 45
Scores on a scale | 3.5 (0.58) | 1.2 (0.61)
Statistical Analysis 1: Comparison: D9421-C 9mg + Mesalazine Placebo vs Mesalazine 3g + D9421-C Placebo; Test type: Superiority or Other; LS mean difference between group = 2.4, 90% CI 2-sided [0.96 to 3.76], Standard Error of Mean 0.84 — [estimate comment as in outcome 4, analysis 1]

27. Secondary Outcome: Change in IBDQ Scores From Baseline to Weeks 10 - Systemic Symptom
Description: as for outcome 16
Time Frame: 10 Week
Population: as for outcome 19
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | D9421-C 9mg + Mesalazine Placebo | Mesalazine 3g + D9421-C Placebo
Number analyzed (Participants) | 50 | 45
Scores on a scale | 3.8 (0.64) | 1.2 (0.62)
Statistical Analysis 1: Comparison: D9421-C 9mg + Mesalazine Placebo vs Mesalazine 3g + D9421-C Placebo; Test type: Superiority or Other; LS mean difference between group = 2.6, 90% CI 2-sided [1.15 to 4.09], Standard Error of Mean 0.89 — [estimate comment as in outcome 4, analysis 1]

28. Secondary Outcome: Change in IBDQ Scores From Baseline to Weeks 2 - Emotional Function
Description: as for outcome 16
Time Frame: 2 Week
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | D9421-C 9mg + Mesalazine Placebo | Mesalazine 3g + D9421-C Placebo
Number analyzed (Participants) | 56 | 54
Scores on a scale | 5.1 (1.00) | 1.3 (1.00)
Statistical Analysis 1: Comparison: D9421-C 9mg + Mesalazine Placebo vs Mesalazine 3g + D9421-C Placebo; Test type: Superiority or Other; LS mean difference between group = 3.8, 90% CI 2-sided [1.44 to 6.19], Standard Error of Mean 1.43 — [estimate comment as in outcome 4, analysis 1]

29. Secondary Outcome: Change in IBDQ Scores From Baseline to Weeks 4 - Emotional Function
Description: as for outcome 16
Time Frame: 4 Week
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | D9421-C 9mg + Mesalazine Placebo | Mesalazine 3g + D9421-C Placebo
Number analyzed (Participants) | 55 | 50
Scores on a scale | 7.0 (1.25) | 2.1 (1.08)
Statistical Analysis 1: Comparison: D9421-C 9mg + Mesalazine Placebo vs Mesalazine 3g + D9421-C Placebo; Test type: Superiority or Other; LS mean difference between group = 4.9, 90% CI 2-sided [2.14 to 7.65], Standard Error of Mean 1.66 — [estimate comment as in outcome 4, analysis 1]

30. Secondary Outcome: Change in IBDQ Scores From Baseline to Weeks 8 - Emotional Function
Description: as for outcome 16
Time Frame: 8 Week
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | D9421-C 9mg + Mesalazine Placebo | Mesalazine 3g + D9421-C Placebo
Number analyzed (Participants) | 51 | 45
Scores on a scale | 5.9 (1.18) | 1.6 (1.31)
Statistical Analysis 1: Comparison: D9421-C 9mg + Mesalazine Placebo vs Mesalazine 3g + D9421-C Placebo; Test type: Superiority or Other; LS mean difference between group = 4.3, 90% CI 2-sided [1.40 to 7.25], Standard Error of Mean 1.76 — [estimate comment as in outcome 4, analysis 1]

31. Secondary Outcome: Change in IBDQ Scores From Baseline to Weeks 10 - Emotional Function
Description: as for outcome 16
Time Frame: 10 Week
Population: as for outcome 19
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | D9421-C 9mg + Mesalazine Placebo | Mesalazine 3g + D9421-C Placebo
Number analyzed (Participants) | 50 | 45
Scores on a scale | 8.0 (1.28) | 1.3 (1.34)
Statistical Analysis 1: Comparison: D9421-C 9mg + Mesalazine Placebo vs Mesalazine 3g + D9421-C Placebo; Test type: Superiority or Other; LS mean difference between group = 6.6, 90% CI 2-sided [3.56 to 9.72], Standard Error of Mean 1.86 — [estimate comment as in outcome 4, analysis 1]

32. Secondary Outcome: Change in IBDQ Scores From Baseline to Weeks 2 - Social Function
Description: as for outcome 16
Time Frame: 2 Week
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | D9421-C 9mg + Mesalazine Placebo | Mesalazine 3g + D9421-C Placebo
Number analyzed (Participants) | 56 | 54
Scores on a scale | 1.9 (0.45) | 0.6 (0.55)
Statistical Analysis 1: Comparison: D9421-C 9mg + Mesalazine Placebo vs Mesalazine 3g + D9421-C Placebo; Test type: Superiority or Other; LS mean difference between group = 1.2, 90% CI 2-sided [0.01 to 2.43], Standard Error of Mean 0.73 — [estimate comment as in outcome 4, analysis 1]

33. Secondary Outcome: Change in IBDQ Scores From Baseline to Weeks 4 - Social Function
Description: as for outcome 16
Time Frame: 4 Week
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | D9421-C 9mg + Mesalazine Placebo | Mesalazine 3g + D9421-C Placebo
Number analyzed (Participants) | 55 | 50
Scores on a scale | 2.5 (0.58) | 0.7 (0.56)
Statistical Analysis 1: Comparison: D9421-C 9mg + Mesalazine Placebo vs Mesalazine 3g + D9421-C Placebo; Test type: Superiority or Other; LS mean difference between group = 1.8, 90% CI 2-sided [0.42 to 3.12], Standard Error of Mean 0.81 — [estimate comment as in outcome 4, analysis 1]

34. Secondary Outcome: Change in IBDQ Scores From Baseline to Weeks 8 - Social Function
Description: as for outcome 16
Time Frame: 8 Week
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | D9421-C 9mg + Mesalazine Placebo | Mesalazine 3g + D9421-C Placebo
Number analyzed (Participants) | 51 | 45
Scores on a scale | 2.3 (0.57) | 0.7 (0.63)
Statistical Analysis 1: Comparison: D9421-C 9mg + Mesalazine Placebo vs Mesalazine 3g + D9421-C Placebo; Test type: Superiority or Other; LS mean difference between group = 1.6, 90% CI 2-sided [0.19 to 3.04], Standard Error of Mean 0.86 — [estimate comment as in outcome 4, analysis 1]

35. Secondary Outcome: Change in IBDQ Scores From Baseline to Weeks 10 - Social Function
Description: as for outcome 16
Time Frame: 10 Week
Population: as for outcome 19
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | D9421-C 9mg + Mesalazine Placebo | Mesalazine 3g + D9421-C Placebo
Number analyzed (Participants) | 50 | 45
Scores on a scale | 2.4 (0.63) | 1.2 (0.56)
Statistical Analysis 1: Comparison: D9421-C 9mg + Mesalazine Placebo vs Mesalazine 3g + D9421-C Placebo; Test type: Superiority or Other; LS mean difference between group = 1.3, 90% CI 2-sided [-0.15 to 2.76], Standard Error of Mean 0.85 — [estimate comment as in outcome 4, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse events collected from the date of signing of informed consent to Visit 6 or withdrawal visit (including the tapering period)
Arm/Group | D9421-C 9mg + Mesalazine Placebo | Mesalazine 3g + D9421-C Placebo
Serious Adverse Events (participants affected / at risk) | 3/56 | 1/56
Other Adverse Events (participants affected / at risk) | 11/56 | 16/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | D9421-C 9mg + Mesalazine Placebo (N=56) | Mesalazine 3g + D9421-C Placebo (N=56)
Ileus (Gastrointestinal disorders) | 1 (1) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | D9421-C 9mg + Mesalazine Placebo (N=56) | Mesalazine 3g + D9421-C Placebo (N=56)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Nasopharyngitis (Infections and infestations) | 6 (6) | 10 (10)
Pharyngitis (Infections and infestations) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 3 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All PIs were prohibited to disclose all information related to this study without AZ approval before this study was completed.